CLINICAL TRIAL: NCT04170907
Title: Randomized Crossover Study Comparing the Pharmacokinetics and Pharmacodynamics of Two Different Nicotine Salt Concentrations and Free-base Nicotine Using an Open Vape Pod System
Brief Title: Pharmacokinetics and Pharmacodynamics of Different Nicotine Salt Concentration Vape System Pods and Free-base Nicotine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: Nicotine PK PD
Record Dates: First submitted 2019-11-12; First posted 2019-11-20 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Nicotine Dependence
Keywords: nicotine; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: Participants will be switched in a within-subject crossover design among the three product types.
Who Masked: Participant, Investigator
Masking Description: Vaping of high and low concentration nicotine salt and free-base nicotine will be double-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nicotine salt 20 mg/mL (Other): Vaping of nicotine salt e-liquids with a nicotine concentration of 20 mg/mL.
  Interventions: Other: standardized vaping protocol
- Nicotine salt 40 mg/mL (Other): Vaping of nicotine salt e-liquids with a nicotine concentration of 40 mg/mL.
  Interventions: Other: standardized vaping protocol
- Free-base nicotine 20 mg/mL (Other): Vaping of free-base nicotine e-liquids with a nicotine concentration of 20 mg/mL.
  Interventions: Other: standardized vaping protocol

INTERVENTIONS:
Other: standardized vaping protocol — The following questionnaires will first be completed: Modified Minnesota Nicotine Withdrawal Scale, Tiffany Questionnaire on Smoking Urges-Brief total (global) craving score, Positive and Negative Affect Schedule. The assigned product will then be given to the participant, and one puff will be taken every 30 seconds (total of 10 puffs). Blood samples will be collected 15 minutes before vaping and 2, 5, 15, 30, 60, 120, and 180 minutes after the last puff. Heart rate and blood pressure will be measured 15 minutes before and 2, 10, 15, 30, 60, 120, and 180 minutes after the last puff. Post-use withdrawal, craving, reward, and satisfaction will be assessed 10 minutes and 1 and 3 hours after the last puff. Respiratory Symptoms will be assessed at baseline and 5 minutes after the last puff. Ten minutes post-use, the direct effects will also be assessed.

SUMMARY:
Comparison of the pharmacokinetics and pharmacodynamics of two different nicotine salt concentrations and free-base nicotine using an open vape pod system

DETAILED DESCRIPTION:
On each study day, one puff will be taken with the assigned product every 30 seconds (total of 10 puffs). Blood samples will be collected to measure nicotine 15 minutes before vaping and 2, 5, 15, 30, 60, 120, and 180 minutes after the last puff. Heart rate and blood pressure will be measured 15 minutes before and 2, 10, 15, 30, 60, 120, and 180 minutes after the last puff. Post-use withdrawal, craving, reward, and satisfaction will be assessed 10 minutes and 1 and 3 hours after the last puff using the modified Minnesota Nicotine Withdrawal Scale (MNWS), the Tiffany Questionnaire on Smoking Urges (QSU), and the Positive and Negative Affect Schedule (PANAS) questionnaires. Respiratory symptoms will be assessed at baseline and 5 minutes after the last puff. Ten minutes post-use, the direct effects of the assigned product (e.g. satisfying, calming, pleasant, vape another one right now) will also be assessed using visual analog scales.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, age 18 or older at screening, who have used electronic cigarettes and/or smoked at least 5 cigarettes per day in the past 30 days
* Saliva cotinine of > 50 ng/mL at screening
* No clinically significant findings on the physical examination at screening
* Ability to communicate well with the investigator and to understand and comply with the requirements of the study
* Women of child-bearing age: willingness of using a reliable contraception method during the study
* Signed informed consent

Exclusion Criteria:

* Known hypersensitivity/allergy to a content of the e-liquid
* Pregnancy or breast feeding
* BMI < 18 or > 28 kg/m2 at screening
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to screening
* Loss of ≥ 250 ml of blood within 3 months prior to screening, including blood donation
* Treatment with an investigational drug within 30 days prior to screening
* Treatment with prescribed or over-the-counter (OTC) medications with potential influence on CYP2A6 function within 1 week prior to screening (with the exception of contraception)
* History or clinical evidence of any disease (e.g. gastrointestinal tract-disease) and/or existence of any surgical or medical condition, which in the opinion of the investigator might interfere with the absorption, distribution, metabolism or excretion of the study drugs, or which might increase the risk for toxicity
* Legal incapacity or limited legal capacity at screening
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Nicotine Peak Plasma Concentration (Cmax) | Blood samples collection: 15 minutes before and 2, 5, 15, 30, 60, 120, and 180 minutes after the last puff
  Comparison of nicotine Cmax between groups

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | Blood samples collection: 15 minutes before and 2, 5, 15, 30, 60, 120, and 180 minutes after the last puff
  Comparison of the nicotine AUC between groups
Time at which the Cmax is observed (Tmax) | Blood samples collection: 15 minutes before and 2, 5, 15, 30, 60, 120, and 180 minutes after the last puff
  Comparison of the nicotine Tmax between groups
Elimination half-life (t1/2) | Blood samples collection: 15 minutes before and 2, 5, 15, 30, 60, 120, and 180 minutes after the last puff
  Comparison of t1/2 between groups
Genotyping of the hepatic cytochrome P450 enzyme CYP2A6 | Blood sample collection during first session
  CYP2A6 genotype (allele variants)
Nicotine metabolite ratio (NMR) | Assessed at screening visit
  Nicotine clearance assessed using 3'-hydroxycotinine/cotinine ratios
Modified Minnesota Nicotine Withdrawal Scale (MNWS) | Baseline, 10 minutes and 1 and 3 hours after the last puff
  Excluding items relating to sleep disturbance and constipation, including eight items (angry/irritable/frustrated, anxious/nervous, depressed mood/sad, desire or craving to smoke, difficulty concentrating, increased appetite/hungry, restless and impatient), rated on a 0=none to 4=severe scale
Tiffany Questionnaire on Smoking Urges-Brief (QSU) total (global) craving score | Baseline, 10 minutes and 1 and 3 hours after the last puff
  Mean of ten items, rated on a 1=strongly disagree to 7=strongly agree scale
Positive and Negative Affect Schedule (PANAS) | Baseline, 10 minutes and 1 and 3 hours after the last puff
  Including items assigned as Positive or Negative Affect (each score is the sum of ten items, rated on a 1=very slightly/not at all to 5=extremely scale)
Respiratory symptoms | At baseline and 5 minutes after the last puff
  Yes/no: shortness of breath, wheezing, cough, phlegm
Direct effects | Ten minutes post-use
  E.g. satisfying, calming, pleasant, vape another one right now, assessed using visual analog scales (0-100 mm) with a single word scored from left (not at all) to right (extremely)
Heart rate | 15 minutes before and 2, 10, 15, 30, 60, 120, and 180 minutes after the last puff
  Heart rate measurements (bpm)
Systolic blood pressure | 15 minutes before and 2, 10, 15, 30, 60, 120, and 180 minutes after the last puff
  Systolic blood pressure measurements (mmHg)
Diastolic blood pressure | 15 minutes before and 2, 10, 15, 30, 60, 120, and 180 minutes after the last puff
  Diastolic blood pressure measurements (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Evangelia Liakoni, MD, Principal Investigator — Sponsor: Inselspital, Bern University Hospital
Locations (1):
- Inselspital, University Hospital Bern, Bern, Canton of Bern, Switzerland